CLINICAL TRIAL: NCT06547749
Title: Vitamin D Supplementation in Critically Ill Children With Respiratory Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Hassan Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: Vitamin D supplementation
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Vitamin D Supplementation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate the role of vitamin D supplementation in critically ill children with respiratory diseases regarding their outcome.

DETAILED DESCRIPTION:
Vitamin D is involved in the process of immunomodulation, especially in the context of autoimmunity . Vitamin D has multiple pharmacological effects, such as alleviating the inflammatory response, promoting phagocytosis, and inducing lymphocyte proliferation . previous studies have demonstrated that patients with lower serum vitamin D levels had a longer length of hospital stay and might have an independent relationship with the duration of mechanical ventilation (MV) in critically ill children

.

Approved Vitamin D Supplementation Regimens:

The recommended daily allowance (RDA) or adequate intake (AI) suggested by the Institute of Medicine (IOM) and supported by Health Canada are 400 IU for infants and 600 IU for older children.

Approved High-Dose Regimens:

In addition to RDA, the IOM provides a higher age-specific dose called the tolerable upper intake level (UL), which ranges from 1,000 to 4,000 IU.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients admitted in PICU with respiratory disease with age from 1month to 16 years.

Exclusion Criteria:

* Patients admitted in PICU due to causes rather than respiratory disease.

Ages: 1 Month to 16 Years | Sex: All
Age Groups: Child
Study Population: pediatric patients admitted in PICU with respiratory disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | Baseline
  How long the patient will stay in Hospital
Ventilator free day | Baseline
  How long is the free days

REFERENCES:
- [Background] Triantos C, Aggeletopoulou I, Mantzaris GJ, Mouzaki A. Molecular basis of vitamin D action in inflammatory bowel disease. Autoimmun Rev. 2022 Aug;21(8):103136. doi: 10.1016/j.autrev.2022.103136. Epub 2022 Jul 2. PMID 35792343
- [Background] Vanichkulbodee A, Romposra M, Inboriboon PC, Trongtrakul K. Effects of vitamin D insufficiency on sepsis severity and risk of hospitalisation in emergency department patients: a cross-sectional study. BMJ Open. 2023 Jan 17;13(1):e064985. doi: 10.1136/bmjopen-2022-064985. PMID 36653058
- [Background] Han JE, Jones JL, Tangpricha V, Brown MA, Brown LAS, Hao L, Hebbar G, Lee MJ, Liu S, Ziegler TR, Martin GS. High Dose Vitamin D Administration in Ventilated Intensive Care Unit Patients: A Pilot Double Blind Randomized Controlled Trial. J Clin Transl Endocrinol. 2016 Jun;4:59-65. doi: 10.1016/j.jcte.2016.04.004. Epub 2016 May 5. PMID 27419080
- [Background] He M, Cao T, Wang J, Wang C, Wang Z, Abdelrahim MEA. Vitamin D deficiency relation to sepsis, paediatric risk of mortality III score, need for ventilation support, length of hospital stay, and duration of mechanical ventilation in critically ill children: A meta-analysis. Int J Clin Pract. 2021 Apr;75(4):e13908. doi: 10.1111/ijcp.13908. Epub 2020 Dec 20. PMID 33280208
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827